CLINICAL TRIAL: NCT01067768
Title: Reduction of Catheter-associated Urinary Tract Infection With a Daily Nursing Review of the Indication. Randomized Controlled Trial
Brief Title: Reduction of Catheter-associated Urinary Tract Infection With a Daily Nursing Review of the Indication
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital Pablo Tobón Uribe (Other)
Responsible Party: Principal Investigator, Maria Victoria Restrepo, MD, MSc, Hospital Pablo Tobón Uribe
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 5100-66592
Record Dates: First submitted 2010-02-10; First posted 2010-02-12 (Estimated); Results first posted 2011-08-04 (Estimated); Last update posted 2019-03-05 (Actual); Status verified 2019-02

CONDITIONS: Urinary Tract Infections; Urinary Tract; Accessory
Keywords: Urinary Tract Infections; Catheter-associated urinary tract infections; Prevention and control; Controlled clinical trial
MeSH Terms: conditions — Urinary Tract Infections

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Daily review (Experimental): In the intervention group a nurse reviewed daily, by using a checklist designed for this study, the indications and pertinence of the catheter. If it was not indicated she asked the doctor to order the removal of the catheter, but the doctor would make the final decision.
  Interventions: Other: Daily review
- Routine care (No Intervention): In the control group, the attending team would remove the catheter as routine, without any suggestion by the research protocol.

INTERVENTIONS:
Other: Daily review — Daily nursing review of the urinary catheter´s indication. If the patient meets at least one of the entries to stay with bladder catheter, the nurse will record collection in the format but will not contact the health team. If there aren´t indication in the medical record, she contacts at the attending physician and said: "Doctor, I didn´t find record in the history of the indication of the urinary catheter, can we withdraw?. If the physician reported the indication, will be recorded in the format without additional comments.
  The attending physician decides withdraw or no withdraw the urinary catheter
  Other Names: Review for indication
  Arms: Daily review

SUMMARY:
The purpose of this study is to determine whether the daily nurse review of the indication of the urinary catheter compared to the everyday care of the working staff is effective to reduce the rate of catheter-associated urinary tract infection in adults hospitalized.

DETAILED DESCRIPTION:
Healthcare-associated infection (HAI)in hospitalized patients are very frequent, especially the catheter-associated urinary tract infection, which prolongs the hospital stay and costs, and is about 3 times more likely to die during hospitalization than patients not infected.

The measures of aseptic insertion and closed systems of collection, as well as the rational use of the probe reduce the risk for infection.

A checklist that contains the agreed indications of catheter, related to obstruction, incontinence, skin lesions in sacral region, monitoring or surgical procedures allows the daily review of the indication of the probe. If the patient doesn´t meet at least one of the criteria, should be recommended the withdrawal of the catheter.

ELIGIBILITY:
Inclusion Criteria:

* Inpatient with a permanent urinary catheter (balloon catheter)
* Urinary catheter placed in the hospitalization (previous day) or at admission

Exclusion Criteria:

* Urinary tract infection diagnosis at time of the insertion
* Spinal cord injury or neurogenic bladder at admission

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1209 (Actual)
Dates: Start 2009-11; Primary Completion 2010-09 (Actual); Study Completion 2010-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: María V Restrepo, Dr., Principal Investigator — Hospital Pablo Tobón Uribe
Locations (1):
- Hospital Pablo Tobon Uribe, Medellín, Antioquia, Colombia

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Adult patients hospitalized with indwelling urinary catheters at a tertiary care, 300-bed, teaching hospital in Colombia- South America, were recruitment between November 2009 and May 2010.
Pre-assignment Details: 1.325 patients were assessed for eligibility. 143 were excluded (98 urinary infection and 45 spinal cord injury).
Groups:
- Control Group: In the control group, the attending team would remove the catheter as routine, without any suggestion by the research protocol.
Period: Overall Study
Arm/Group | Daily Review | Control Group
Started | 604 | 605
Completed | 604 | 605
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Daily Review | Control Group | Total
Number analyzed (Participants) | 604 | 605 | 1209
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 55 [38 to 69] | 56 [37 to 69] | 55.5 [37 to 69]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 250 | 253 | 503
  Male | 354 | 352 | 706
Diabetes [Number; unit: participants] — Diabetes mellitus registered as a personal history or diagnosed on admission
  participants
    Yes | 88 | 84 | 172
    No | 516 | 521 | 1037
Kidney failure [Number; unit: participants] — Creatinine greater than 2 mg/dL at any time during hospitalization
  participants
    Yes | 104 | 94 | 198
    No | 500 | 511 | 1011
Indication of catheter [Number; unit: participants]
  Obstruction | 28 | 19 | 47
  Incontinence | 3 | 0 | 3
  Monitoring | 268 | 269 | 537
  Procedures | 303 | 316 | 619
  None | 2 | 1 | 3
Unit placement [Number; unit: participants] — Site of insertion of the catheter
  participants
    Emergency | 175 | 167 | 342
    Critical care | 67 | 67 | 134
    Surgery | 271 | 282 | 553
    General room | 34 | 24 | 58
    Before admission | 49 | 49 | 98
    Another | 8 | 16 | 24

OUTCOME MEASURES:

1. Primary Outcome: Rate of Catheter-associated Urinary Tract Infection
Time Frame: Until 7 days after the withdrawal of the catheter or at discharge (whichever comes first)
Population: Analysis by intention to treat
Measure: Number (95% Confidence Interval); unit: infections per 1000 days
Groups:
- Daily Review: Daily monitoring of catheter indication
Arm/Group | Daily Review | Control Group
Number analyzed (Participants) | 604 | 605
infections per 1000 days | 10 [6.58 to 14.02] | 12 [8.85 to 16.34]
Statistical Analysis 1: Comparison: Daily Review vs Control Group; The sample size was calculated for the primary outcome. An infection rate 15 per 1,000 urinary catheter days in the control group and an expected reduction in the intervention group 40% clinically important effect. Mapping one to one, 5% alpha error and beta error 20%; Test type: Superiority or Other; Risk Ratio (RR) = 0.81, 95% CI 2-sided [0.50 to 1.3] — The primary outcome analysis was performed using relative risk (RR) between the rate of urinary tract infection per 1,000 days of exposure of the test subjects to intervention and that of patients undergoing routine care

2. Secondary Outcome: Catheter Days
Description: The duration of catheterization
Time Frame: withdrawal of the catheter
Population: Analysis by intention to treat
Measure: Median (Inter-Quartile Range); unit: Days
Arm/Group | Daily Review | Control Group
Number analyzed (Participants) | 604 | 605
Days | 2 [1 to 5] | 3 [1 to 6]
Statistical Analysis 1: Comparison: Daily Review vs Control Group; Null hypothesis: On average catheterization are the same in patients with daily review of the indication and control group patients; Test type: Superiority or Other; p = 0.016, Wilcoxon (Mann-Whitney) — The difference between groups was evaluated with a U test Mann Whitney. The difference was statistically significant with p values less than 0.05

ADVERSE EVENTS:
Arm/Group | Daily Review | Control Group
Serious Adverse Events (participants affected / at risk) | 0/604 | 0/605
Other Adverse Events (participants affected / at risk) | 0/604 | 0/605

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes